CLINICAL TRIAL: NCT04816162
Title: Ketofol vs Dexmedetomidine for Preventing Post-operative Delirium in Elderly Patients Undergoing Intestinal Obstruction Surgeries. A Randomized Controlled Study
Brief Title: Ketofol for Preventing Postoperative Delirium in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6704/10-3-2021
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Delirium on Emergence
Keywords: ketofol; dexmedetomidine; post operative delirium; elderly patients
MeSH Terms: conditions — Emergence Delirium | interventions — Ketamine; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: A computer-generated table will be used to divide patients equally into three study groups
  * In group C (control group):21 ml of normal saline 0.9% will be I.V infused at a rate of 0.3-0.4 mg/kg/h to the patient.
  * In group K: ketofol (a mixture of ketamine and propofol will be prepared in a ratio of (1:4) respectively), will be I.V infused at a rate of 0.3-0.4 mg/kg/h to the patient.
  * In group D: adding dexmedetomidine 2 ml (200 µg) to 19 ml of 0.9% normal saline to start I.V infusion to the patient
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blinded(participants and outcome assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): 21 ml of normal saline 0.9% will be I.V continuously infused fifteen minutes after induction of anesthesia up to two hours postoperatively.
  Interventions: Other: normal saline
- ketofol group (Active Comparator): 21 ml of a mixture of (ketamine and propofol) will be I.V continuously infused fifteen minutes after induction of anesthesia up to two hours postoperatively
  Interventions: Drug: ketofol
- dexmedetomidine group (Active Comparator): 21 ml of a mixture of (dexmedetomidine diluted with normal saline 0.9%) will be I.V continuously infused fifteen minutes after induction of anesthesia up to two hours postoperatively
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: ketofol — prepared in a ratio of (1:4) respectively), where 1ml of ketamine will be added to 20 ml of propofol in a syringe pump
  Other Names: a mixture of propofol and ketamine
  Arms: ketofol group
Drug: dexmedetomidine — 2 ml (200 µg) of dexmedetomidine added to 0.9% normal saline in a syringe pump
  Other Names: precedex
  Arms: dexmedetomidine group
Other: normal saline — normal saline 0.9% in a syringe pump
  Arms: Control group

SUMMARY:
* Delirium is a cognitive disturbance characterized by acute and fluctuating impairment in attention and awareness. Although its incidence in the general surgical population is 2-3%, it has been reported to occur in up to 10-80% of high-risk patient groups. In addition, the occurrence of postoperative delirium is associated with considerably raised morbidity and mortality and increased healthcare resource expenditure.
* In the general patient population, no prophylactic pharmacologic treatment has shown widespread effectiveness in preventing delirium. Several studies have failed to find a magic pharmacologic bullet for preventing delirium-ketamine, haloperidol, propofol, antipsychotic and benzodiazepine drugs have recently tested without a clear result of its effectiveness.
* Dexmedetomidine is an attractive pharmacologic option because of its biological plausibility in modifying several known contributors to delirium.
* Up to investigators' knowledge, there is no study done to compare the effect of infusion of dexmedetomidine and ketofol mixture as prophylactic agents for high-risk patients as elderly patients who undergoing high-risk surgery such as intestinal obstruction surgery against postoperative delirium occurrence.

DETAILED DESCRIPTION:
Small bowel obstruction (SBO) is one of the most frequent causes of general emergency surgery in elderly patients, approximately 10-12% of adult patients above 65 years presenting with acute abdominal pain at the emergency department (ED) is diagnosed as SBO. Small bowel obstruction is complicated with dehydration, malnutrition, electrolyte and acid-base disturbance, as well as insertion of many catheters as nasogastric tube, triple-lumen tube, and foley's catheter, besides multiple drugs intake due to the associated comorbidities; all of these factors increase the risk of developing POD ].

Delirium is defined as acute onset of fluctuating disturbance of consciousness with reduced ability to focus, alteration of attention, perceptual abnormalities, circadian disruption, a decline in cognitive function (orientation, memory speech, thinking), and psychomotor disturbances. POD commonly occurs between postoperative days 2-5, and it may be hypoactive, hyperactive, or mixed, based on psychomotor clinical features. The incidence rate of postoperative delirium(POD) varies between 9% and 87% in elderly patients, depending on the patients' population and degree of operative stress.

Postoperative delirium develops in the elderly due to multiple risk factors that can be separated into patient-related and operation-related risk factors. Established patient-specific risk factors include pre-existing dementia (appears to be the strongest predictor for the occurrence of POD), older age, functional impairment, greater co-morbidities, and psychopathological symptoms. Operation-specific risk factors for POD are based on the degree of operative stress, any type of iatrogenic event including medication adverse effects (Common drugs that may precipitate delirium in the elderly include antihistamines, anticholinergics, chemotherapeutic agents, dopamine agonists, benzodiazepines, opioid analgesics, steroids, and psychostimulants), physical restraint, urinary catheterization, hospital-acquired infection, dehydration and malnutrition, and admission to the intensive care unit (ICU). The risk factors for developing POD are additive therefore, recognizing those with multiple risk factors should trigger environmental and supportive measures implementation that have been proven to prevent the onset and shorten the duration of POD because POD is associated with poor outcomes such as functional decline, longer hospitalization, greater costs, a greater need for rehabilitation and home healthcare services after discharge and higher mortality.

Ketofol which is a mixture of ketamine and propofol gains increasing interest as an agent for procedural sedation and analgesia for producing a more stable hemodynamic and respiratory profile as Ketamine and propofol appear to counter each other's adverse effects; sympathomimetic effects of ketamine and dose-dependent hypotension and respiratory depression of propofol. Ketofol has been used in different mixed ratios (1:1-1:10) and has proven effective in reducing postoperative agitation in children in several studies as well.

Dexmedetomidine, a highly selective alpha-2 adrenoreceptor (α2) agonist, has been widely used in surgical patients and has positive sedation, anti-anxiety, and analgesic effects. The mechanism of action of dexmedetomidine is unique compared with traditionally administered sedative agents due to its lack of activity at the gamma-aminobutyric acid (GABA) receptor and missing anticholinergic activity.1that may contribute to pathophysiological explanations of the development of delirium 'neurotransmitter hypothesis' and include dysfunction of cholinergic transmission.

The investigators hypothesized that administration of ketofol following induction of general anesthesia, would reduce the incidence of emergence delirium and postoperative delirium, and has a comparable effect to dexmedetomidine on investigators' groups of high-risk elderly patients undergoing urgent exploration of intestinal obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age ≥ 60 years old.
* American society of anesthesia (ASA) (II-III).
* Gender: males &females
* BMI < 35kg/m2.
* able to communicate verbally.
* Scheduled for exploration surgery for intestinal obstruction under general anesthesia of at least 60 min duration

Exclusion Criteria:

* Patient refusal.
* Patients with delirium prior to surgery.
* Patients with drug misuse history or taking anti-psychotic drugs.
* Previous hospitalization within 3 months.
* Legal blindness, severe deafness.
* History of Acute cerebrovascular conditions; stroke or transient ischemic attack.
* Patients who could not be prepared with proper fluid resuscitation, electrolyte and acid-base correction prior to surgery.
* Patients who could be discharged from the intensive care unit (ICU) within two days.
* Patients with a known history of allergy to study drugs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
incidence of post operative delirium | up to first three postoperative days
  Patients will be assessed for postoperative delirium using Confusion Assessment Method (CAM), or the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)

SECONDARY OUTCOMES:
changes of pain assessment | 30 minutes, 1 hour, 2, 4, 18, 12, 24 hours postoperatively
  Visual analogue scale
changes of hemodynamics | immediately prior to surgery, intraoperative (after starting infusion of study drug, then every 10 minute till end of surgery), later on they will be measured every 15 min postoperatively up to two hours postoperatively
  by non invasive blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E Abd Ellatif, MD, Principal Investigator — faculty of human medicine,zagazig university
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Alsharqia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: planned after the completion of the study and publication
Access Criteria: contact with principal investigator

REFERENCES:
- [Background] Spangler R, Van Pham T, Khoujah D, Martinez JP. Abdominal emergencies in the geriatric patient. Int J Emerg Med. 2014 Oct 21;7:43. doi: 10.1186/s12245-014-0043-2. eCollection 2014. PMID 25635203
- [Background] Ozturk E, van Iersel M, Stommel MM, Schoon Y, Ten Broek RR, van Goor H. Small bowel obstruction in the elderly: a plea for comprehensive acute geriatric care. World J Emerg Surg. 2018 Oct 20;13:48. doi: 10.1186/s13017-018-0208-z. eCollection 2018. PMID 30377439
- [Background] Dale O, Somogyi AA, Li Y, Sullivan T, Shavit Y. Does intraoperative ketamine attenuate inflammatory reactivity following surgery? A systematic review and meta-analysis. Anesth Analg. 2012 Oct;115(4):934-43. doi: 10.1213/ANE.0b013e3182662e30. Epub 2012 Jul 23. PMID 22826531
- [Background] Maldonado JR, Wysong A, van der Starre PJ, Block T, Miller C, Reitz BA. Dexmedetomidine and the reduction of postoperative delirium after cardiac surgery. Psychosomatics. 2009 May-Jun;50(3):206-17. doi: 10.1176/appi.psy.50.3.206. PMID 19567759
- [Background] Li WX, Luo RY, Chen C, Li X, Ao JS, Liu Y, Yin YQ. Effects of propofol, dexmedetomidine, and midazolam on postoperative cognitive dysfunction in elderly patients: a randomized controlled preliminary trial. Chin Med J (Engl). 2019 Feb;132(4):437-445. doi: 10.1097/CM9.0000000000000098. PMID 30707179
- [Background] Smischney NJ, Hoskote SS, Gallo de Moraes A, Racedo Africano CJ, Carrera PM, Tedja R, Pannu JK, Hassebroek EC, Reddy DR, Hinds RF, Thakur L. Ketamine/propofol admixture (ketofol) at induction in the critically ill against etomidate (KEEP PACE trial): study protocol for a randomized controlled trial. Trials. 2015 Apr 21;16:177. doi: 10.1186/s13063-015-0687-0. PMID 25909406
- [Derived] Abd Ellatif SE, Mowafy SMS, Shahin MA. Ketofol versus Dexmedetomidine for preventing postoperative delirium in elderly patients undergoing intestinal obstruction surgeries: a randomized controlled study. BMC Anesthesiol. 2024 Jan 2;24(1):1. doi: 10.1186/s12871-023-02378-5. PMID 38166598